CLINICAL TRIAL: NCT00919243
Title: Prednisone Versus Allopurinol for Symptomatic Heart Failure Patients With Hyperuricemia
Brief Title: Prednisone for Heart Failure Patients With Hyperuricemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Professor, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hebmu 08-12
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2009-06

CONDITIONS: Heart Failure; Hyperuricemia
Keywords: prednisone; allopurinol; heart failure; hyperuricemia
MeSH Terms: conditions — Heart Failure; Hyperuricemia | interventions — Prednisone; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prednisone (Experimental)
  Interventions: Drug: prednisone
- allopurinol (Active Comparator)
  Interventions: Drug: allopurinol

INTERVENTIONS:
Drug: prednisone — 1 mg/kg/day with a maximum dose of 60 mg/day given orally
  Arms: prednisone
Drug: allopurinol — allopurinol, the dose of allopurinol is adjusted by patients' renal function, and with a maximum dose of 300mg/day.
  Arms: allopurinol

SUMMARY:
Hyperuricemia is a very common finding in patients with heart failure. It is usually related to diuretic use and deteriorated renal function. The recently evidence showed that uric acid (UA) lowering therapy may improve clinical status in symptomatic heart failure patients with hyperuricemia. In their clinical practice, the investigators found that glucocorticoids could dramatically lower UA while improving renal function. Thus the investigators design this randomized head to head study to test our hypothesis that prednisone have the same efficacy to allopurinol on lowering UA and could improve renal function at the same time.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* NYHA Class III-IV
* EF =< 40%
* Uric acid => 9.5 mg/dL

Exclusion Criteria:

* Acute gouty arthritis
* Any condition (other than CHF) that could limit the use of prednisone or allopurinol
* Any concurrent disease likely to limit life expectancy.
* Active myocarditis, or an obstructive or restrictive cardiomyopathy
* Heart Attack, Stroke, Unstable Angina or Cardiac surgery within previous 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in uric acid level | 4 weeks

SECONDARY OUTCOMES:
Change from baseline in creatinine clearance rate | 4 weeks
Daily urine volume | 4 weeks
Body weight | 4 weeks
patient assessed dyspnea and physician assessed global clinical status | 4 weeks
6-minute walking distance | 4 weeks
NYHA functional class | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kunshen Liu, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Liu C, Zhao Q, Zhen Y, Gao Y, Tian L, Wang L, Ji L, Liu G, Ji Z, Liu K. Prednisone in Uric Acid lowering in Symptomatic Heart Failure Patients With Hyperuricemia (PUSH-PATH) study. Can J Cardiol. 2013 Sep;29(9):1048-54. doi: 10.1016/j.cjca.2012.11.008. Epub 2013 Feb 6. PMID 23395281